CLINICAL TRIAL: NCT05698927
Title: Can Erector Spinae Plane Block Replace Intrathecal Morphine in Cesarean Section? a Prospective Randomized Controlled Study on Opioid Consumption
Brief Title: Analgesic Effects of Intrathecal Morphine and Bilateral Erector Spina Plane Block in Elective Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MarmaraMedical
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Opioid Use; Postoperative Pain
Keywords: postoperative pain; opioid consumption; erector spinae plane block; intrathecal morphine
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrathecal Morphine Group (Active Comparator): Bilateral Erector Spinae Plane Block (with %0.25 bupivacaine, 20 ml for each side) and intravenous tramadol via Patient Controlled Analgesia device (5 mg/ml tramadol, bolus dose: 1ml, lock time: 20 minutes)
  Comparing postoperative pain and opioid consumption in groups
  Interventions: Procedure: Erector Spinae Plane Block (bilaterally, via 20ml % 0.25 bupivacain) and Intrathecal Morphine (100 mcg)
- Bilateral Erector Spinae Plane Block Group (Active Comparator): Intrathecal morphine (100mcg) and intravenous tramadol via Patient Controlled Analgesia device (5 mg/ml tramadol, bolus dose: 1ml, lock time: 20 minutes) Comparing postoperative pain and opioid consumption in groups
  Interventions: Procedure: Erector Spinae Plane Block (bilaterally, via 20ml % 0.25 bupivacain) and Intrathecal Morphine (100 mcg)

INTERVENTIONS:
Procedure: Erector Spinae Plane Block (bilaterally, via 20ml % 0.25 bupivacain) and Intrathecal Morphine (100 mcg) — Comparison of the postoperative opioid consumptions between Erector Spinae Plane Block (bilaterally, via 20ml % 0.25 bupivacain) and Intrathecal Morphine (100 mcg)

SUMMARY:
Cesarean section cause severe pain due to surgical incision, abdominal wall retraction and visceral organ movements. Cesarean section can be performed with general anesthesia, spinal anesthesia, epidural anesthesia and combined spinal epidural anesthesia methods.

Because of the possibility of aspiration pneumonia in pregnant women are under general anesthesia, the awareness of anesthesia in the mother during the operation due to insufficient anesthesia, unsuccessful intubation, respiratory complications in the mother and newborn and low APGAR scores, regional anesthesia is superior to general anesthesia in elective cesarean section operations.

Spinal anesthesia, abdominal wall blocks such as erector spinae plane block, parenteral and intrathecal opioids may be used for postoperative analgesia in cesarean section operations.

Intrathecal morphine can cause postoperative nausea-vomiting, itching, respiratory depression. Erector spina plane block can provide effective pain control and reduce opioid consumption.

The primary implication of this study is to compare postoperative pain scores and opioid consumption on elective cesarean section patients under spinal anesthesia with intrathecal morphine or erector spina block in addition to spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 40 years old, ASA (American Society of Anesthesiologists) score I-II, undergoing elective cesarean section

Exclusion Criteria:

* Emergency cesarean section
* The patients with major hepatic, cardiovascular or renal disease
* The patients for whom spinal anesthesia is contraindicated
* The patients who is allergic to any drugs that we use for this study
* Patients who declined to participate in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption | 24 hours
  Comparing opioid (tramadol) consumption via intravenous Patient Controlled Analgesia (PCA) device

SECONDARY OUTCOMES:
Pain Scores | 24 hours
  In a Numerical Rating Scale (NRS), patients are asked to choose the number between 0 and 10, that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas ten represents 'the worst pain ever possible'
Rescue analgesia | 24 hours
  when the patient's NRS score ≥ 4, diclofenac 75 mg intramuscular is given
Side effects of medications | 24 hours
  Intravenous and intrathecal opioids can cause nausea-vomiting, itching, respirator depression

OTHER OUTCOMES:
Participant satisfaction | 24 hours
  Comparing pain with numeric rating scale (NRS) In a Numerical Rating Scale (NRS), patients are asked to choose the number between 0 and 10, that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas ten represents 'the worst pain ever possible'
Apgar scores of newborns | 1st and 5th minute after the delivery.
  APGAR (Activity, Pulse, Grimace, Appearance, Respiration) score is a measure of the physical condition of a newborn infant. It is obtained by adding points (2, 1, or 0) for heart rate, respiratory effort, muscle tone, response to stimulation, and skin coloration; a score of 10 represents the best possible condition. It may be effected by intravenous or intrathecal opioids that is given to mother.

CONTACTS AND LOCATIONS:
Overall Officials: Beliz Bilgili, Study Chair — Marmara University
Locations (2):
- Turkey (Türkiye) (2):
  - Marmara University School of Medicine, Istanbul
  - Marmara University, Istanbul